CLINICAL TRIAL: NCT05175807
Title: Application of a Telemedicine Brief Mindfulness Intervention in Post-COVID-19: a Pilot Randomized and Controlled Trial
Brief Title: A Telemedicine Brief Mindfulness Intervention in Post-COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Paolo Banfi, MD, Chief of the Cardio-Respiratory Rehabilitation, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FDG_MNF-COVID19
Record Dates: First submitted 2021-04-22; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Post COVID-19
Keywords: Post COVID-19; Mindfulness; Randomized Controlled Trial; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Group_1 (Experimental): The intervention will be characterized by be based on Mindfulness exercises (e.g. body scan, gentle yoga, sitting, grounding and walking meditation), relaxation techniques and cognitive rehabilitation exercises. walking), relaxation techniques and cognitive rehabilitation exercises. The objective is to provide specific practical skills to learn how to deal with difficult and/or stressful situations managing emotions and intercurrent thoughts. The intervention is proposed to last for a total of 5-6 sessions lasting 45 minutes each, two sessions per week, for a three-week commitment. In addition, between sessions, reflection materials, readings or exercises will be offered. The intervention will be conducted in telemedicine by a Psychologist, who has experience in conducting these interventions and who receives regular supervision. The sessions will be conducted through special platform and audio-recorded to ensure the reliability of the data collected, prior consent.
  Interventions: Other: Mindfulness
- Waiting List Group_2 (No Intervention): In both groups the "usual care" or usual treatment, will consist of the usual daily medical examinations of the department, respiratory and motor physiotherapy sessions. The Group 2, therefore, will not be submitted to other type of treatment outside of that previewed near O.U. for the course of the first three weeks, during which they will be placed on the waiting list. Once the Once the assessment is carried out after 3 weeks, we will proceed to implement the intervention proposed to the Group 1. If the participant has already been discharged from the structure, it will still be possible to proceed with the intervention, since it is online. If the participant has already been discharged from the structure, you can still proceed with the intervention, since this is in telemedicine, in order to promote the continuity hospital-territory.

INTERVENTIONS:
Other: Mindfulness — Mindfulness (e.g., body scan, gentle yoga, sitting, grounding, and walking meditation), relaxation techniques, and cognitive rehabilitation exercises.
  Arms: Mindfulness Group_1

SUMMARY:
Background: Several studies suggest that SARS survivors still presented with high levels of psychological distress overall at 1, 3, 12, and 18 months after hospital discharge. Nonetheless, there are no data available in the literature regarding the implementation of interventions that are psychological interventions, let alone specific ones. In particular, the practice of mindfulness, formalized in the protocols such as Mindfulness Based Stress Reduction (MBSR) and Mindfulness Based Cognitive Therapy (MBCT). Based Cognitive Therapy (MBCT), have proved to be very effective in reducing stress related to chronic conditions and of depression. However, these protocols typically require a high level of engagement for participants, which is why, in the present exploratory study, the investigators opted to evaluate the implementation of a Mindfulness-based protocol that is short and less intense, but which has shown good results on health-related outcomes, even with a single session.

Objectives: In this perspective, it becomes important to detect the presence of psychological distress in those who have contracted COVID-19 and are now undertaking a rehabilitation program, from the perspective of promoting well-being and prevention of possible aggravation if not prolongation of mental suffering in the long term.

Study Design: Randomized and Controlled (RCT), two-arm pilot study with three data captures (baseline=T0, 3 weeks=T1, 3 months=T2).

Participants: People who have previously tested positive for COVID-19, now negative and hospitalized at the IRCCS Santa Maria Nascente of the Fondazione Don Carlo Gnocchi in Milan.

ELIGIBILITY:
Inclusion Criteria:

* Previously positive for COVID-19 and now negative and undergoing treatment Pulmonary rehabilitation;
* Compatibility to participate in the study as judged by the physician;
* Able to provide Informed Consent.

Exclusion Criteria:

* The physician's unfavorable opinion of inclusion in the study because he or she is unable to provide Informed Consent;
* Patients with lung cancer;
* Documented psychiatric disorders;
* Immunodepression;
* Patients with terminal or neurodegenerative diseases (e.g., other forms of cancer, Amyotrophic Lateral Sclerosis (ALS)).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms of Post-Traumatic Stress Disorder (PTSD) | Change from baseline at 3 weeks and at 3 months
  Symptoms of Post-Traumatic Stress Disorder (PTSD) as measured by the Impact of Event Scale (IES) (Horowitz, Wilner, & Alvarez, 1979). The revised version of the Impact of Event Scale (IES-r) has seven additional questions and a scoring range of 0 to 88.
  On this test, scores that exceed 24 can be quite meaningful. High scores have the following associations.

SECONDARY OUTCOMES:
Anxiety 2006), at baseline, 3 weeks, 3 months after recruitment. | Change from baseline at 3 weeks and at 3 months
  Anxiety, detected through the General Anxiety Disorder (GAD-7)(R L Spitzer, K Kroenke, Williams, & Lowe, 2006). The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions.
  GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.
  When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Depression | Change from baseline at 3 weeks and at 3 months
  Depression, detected through the Patient Health Questionnaire (PHQ-9) (Löwe, Kroenke, Herzog, & Gräfe, 2004). Each item is evaluated on a severity scale ranging from 0 to 3 where the respondent is asked to rate how often each symptom occurred over the last 2 weeks (0-not at all; 1-several days; 2-more than half of the days or 3-nearly every day), yielding a total score ranging from 0-27. The respondent is also asked how the identified problems have interfered with work, home and/or social life, however responses to this item are not scored or included in the total score.
  Score interpretation:
  1-4 minimal depression; 5-9 mild depression; 10-14 moderate depression; 15-19 moderately severe depression; and 20-27 severe depression
Psychological distress | Change from baseline at 3 weeks and at 3 months
  Psychological distress, measured by the Perceived Stress Scale (PSS)(Cohen, S., Kamarck, T., & Mermelstein, 1994). PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made from questions 2, 4, 5 and 10 of the PSS 10 item scale.
Counterfactual thinking and peritraumatic emotions of guilt, shame, and fear in relation to the events stressful events | Change from baseline at 3 weeks and at 3 months
  Counterfactual thinking and peritraumatic emotions of guilt, shame, and fear in relation to stressful events stressful events as measured by the State Shame and Guilt Scale-8 (Cavalera, Pepe, Zurloni, Diana, & Realdon, 2017) and the Peritraumatic Perceptions of Fear and life threat (Breiding et al., 2015;Tran & Beck, 2019). Scoring Each scale consists of 5 items: Shame - Items 1, 3, 5, 7, 9 Guilt - Items 2, 4, 6, 8, 10 All items are scored in a positive direction.
Well-being | Change from baseline at 3 weeks and at 3 months
  Well-being, as measured by the Psychological General Well-being Index (PGWBI)(Chassany, Dimenas, Dubois, Wu, & Dupoy, 2004; Grossi & Compare, 2014). The PGWBI global score represents the sum of all items and ranges from 0 to 110. Higher scores indicate greater psychological well-being.
Changes with respect to respiratory function | Change from baseline at 3 weeks and at 3 months
  Changes with respect to respiratory function, as measured by Forced Vital Capacity (CVF), Forced Expiratory Forced Expiratory Volume in 1 Second (VEF1) and Tiffenau's Index (VEF1/CVF)
Changes in arterial blood gas analysis (ABG) | Change from baseline at 3 weeks and at 3 months
  Changes in arterial blood gas analysis (ABG), which measures oxygen tension (PaO2) and that of carbon dioxide (PaCO2)
Changes in oxygen saturation (SpO2) | Change from baseline at 3 weeks and at 3 months
  Changes in oxygen saturation (SpO2)
Change in CBC, ferritin, fibrinogen, creatinine, electrolytes, transaminases, d-dimer values, immunoelectrophoresis, baseline cortisolemia ACTH, CPK, COVID-19-related serological values of IgG and IgM. | Change from baseline at 3 weeks and at 3 months
  Change in CBC, ferritin, fibrinogen, creatinine, electrolytes, transaminases, d-dimer values, immunoelectrophoresis, baseline cortisolemia ACTH, CPK, COVID-19-related serological values of IgG and IgM.
CBC, basal cortisolemia ACTH, CPK | Change from baseline at 3 weeks and at 3 months
  CBC, basal cortisolemia ACTH, CPK

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Santa Maria Nascente, Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cavalera, C., Pepe, A., Zurloni, V., Diana, B., & Realdon, O. (2017). A short version of the state shame and guilt scale (SSGS-8). TPM - Testing, Psychometrics, Methodology in Applied Psychology, 24(1), 99-106. https://doi.org/10.4473/TPM24.1.6
- [Background] Cohen, S., Kamarck, T., & Mermelstein, R. (1994). Perceived Stress Scale. In Measuring stress: A guide for health and social scientists (p. 10).
- [Background] Grossi, E., & Compare, A. (2014). Psychological General Well-Being Index (PGWB). In Encyclopedia of Quality of Life and Well-Being Research. https://doi.org/10.1007/978-94-007-0753-5_2309
- [Background] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Background] Lowe B, Kroenke K, Herzog W, Grafe K. Measuring depression outcome with a brief self-report instrument: sensitivity to change of the Patient Health Questionnaire (PHQ-9). J Affect Disord. 2004 Jul;81(1):61-6. doi: 10.1016/S0165-0327(03)00198-8. PMID 15183601
- [Background] Tran, H. N., & Beck, J. G. (2019). Are Peritraumatic Perceptions of Fear/Life Threat and Posttraumatic Negative Self-Conscious Appraisals/Emotions Differentially Associated with PTSD Symptoms? Cognitive Therapy and Research, 43(1), 272-283.